CLINICAL TRIAL: NCT04439877
Title: Exploring the Relationship Among Dental Caries, Nutritional Habits and Peri-implantitis
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Javi Vilarrasa, Assistant Professor at the Department of Periodontology, Universitat Internacional de Catalunya
Other Study IDs: PER-ECL-2017-08
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Peri-Implantitis; Mucositis; Caries,Dental; Nutrition
MeSH Terms: conditions — Peri-Implantitis; Mucositis; Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Peri-implant disease diagnosis — Diagnosis of peri-implant disease

SUMMARY:
Aim: A study was made of the prevalence, co-occurrence and association among caries, nutritional habits and peri-implant disease, with an analysis of the influence of other patient and implant factors upon peri-implant disease.

Material and methods: The included subjects underwent a clinical examination and were asked to complete a questionnaire. Demographic data and potential lifestyle/behavioral variables were collected. Clinical and radiographic assessment allowed calculation of the decayed, missing and filled teeth (DMFT) index and peri-implant diagnosis. Uni- and multivariate logistic regression analyses were applied to identify predictors of peri-implant disease.

DETAILED DESCRIPTION:
2.1. Study design

The present cross-sectional study was conducted after approval from the local Ethics Committee (Ref. PER-ECL-PER-2017-08) and in accordance with the ethical principles outlined in the Declaration of Helsinki. It is reported according the Strengthening the Reporting of Observational Studies Epidemiology (STROBE) statement recommendations (von Elm et al., 2009). Selected subjects were informed about the aims of the research, and written consent was obtained before starting the study.

2.2. Study population

Patients visiting the Postgraduate Periodontology Clinic of the Faculty of Dentistry of the Universitat Internacional de Catalunya (Barcelona, Spain) from January 2018 to December 2019 were consecutively enrolled in the study by one of the researchers (JV), if they met the criteria addressed later on in the form.

2.3. Data collection

Data collection comprised a patient interview and clinical and radiographic assessment. Initially, a previously trained examiner (MP) interviewed the patients and collected the following data:

* Age (years).
* Gender (female/male).
* Smoking habit: smoker, non-smoker or ex-smoker. In the case of smokers, the total amount of cigarettes per day was categorized as < 10 or more than 10 cigarettes per day.
* Systemic diseases: presence or absence.
* Diabetes mellitus: presence or absence. In the case of diabetic patients, glycemic control was assessed on the basis of a previous blood test.
* Body mass index (BMI): recorded as weight (kg)/ height (m)2.
* Dietary habits: assessed by the Mediterranean Diet Score (MDS) questionnaire (Martínez-González et al., 2012) and classified as low adherence (score ≤ 5), medium adherence (score 6-9) or high adherence (score ≥10).
* Regular sugar consumption: yes or no. Sugar consumers were also asked about their level of sugar intake (low, medium, high).
* Nutrient or vitamin deficiencies: presence or absence.
* Oral dryness: patient perception of dry mouth (presence or absence).
* Educational level (EL): primary and secondary or professional and university.
* Oral hygiene measures: frequency of teeth brushing and interproximal hygiene.
* Supportive periodontal treatment (SPT): regular (≥ 2 times/year) or irregular (< 2 times/year).
* Cause of tooth loss: caries, mobility, caries and mobility, and trauma/fracture.

Any doubts coming from the questionnaire were solved by the examiner. A previously calibrated examiner (LG) conducted the intraoral examination (with a Cohen inter-agreement kappa index > 85%). The exploration was conducted to assess the following parameters:

* Periodontal indexes: full mouth plaque score (FMPS) (O'Leary et al. 1972) and bleeding score (FMBS) (Ainamo & Bay 1975).
* History of periodontitis: assessed radiographically by the presence or absence of bone loss.
* Number of decayed, missing and filled teeth (DMFT) assessed by visual inspection and radiographic assessment following the ICDAS (Pitts & Ekstrand, 2013). All tooth surfaces were examined, but the observations were recorded per tooth.
* Probing pocket depth (PPD) (in mm), bleeding on probing (BoP) (yes/no), suppuration (SUP) (yes/no), keratinized mucosa (KM) (in mm) were all recorded at 6 sites per implant using a PCP UNC 15 probe (Hu-Friedy ®).
* Radiographic bone level (in mm) at mesial and distal to the implant site using the parallel cone technique.
* Implant position (anterior maxilla, anterior mandible, posterior maxilla, posterior mandible).
* Interproximal untreated caries or fillings adjacent to implants: yes/no. If these conditions were present, their location was recorded (mesial, distal or both).

Patients presenting with caries or periodontal or peri-implant disease were referred to the corresponding clinical department within the Universitat Internacional de Catalunya for further evaluation and management.

2.4. Outcome measures

The main outcome measure of the study was the prevalence of dental caries and peri-implant disease.

All other variables obtained from the questionnaire and clinical examination were regarded as secondary outcome measures.

2.5. Sample size calculation

A logit regression model used to associate the outcome diagnosis at the patient level and each exposure variable reached a statistical power of 82.5% in detecting odds ratio (OR) = 2.5 as being significant in the recruited sample (n= 169), assuming a confidence level of 95%. At the implant level, the power was 96.2% under the same previous conditions. Due to the multi-level design, the power had to be corrected. In this regard, assuming a moderate intra-subject correlation (ρ = 0.5), a power of 87.7% was estimated.

2.6. Statistical analysis

A descriptive analysis was carried out, with the calculation of absolute and relative frequencies (categorical variables) and the mean and standard deviation (SD) (continuous variables).

At patient level, simple binary logistic regression models were estimated to study the association between the patient diagnosis (H versus M, and H versus PI) and each of the exposure variables. At implant level, simple binary logistic regression models were estimated using generalized estimating equations (GEEs). The models estimated odds ratio (OR) from the Wald chi-squared statistic. The GEE approach addressed intra-subject dependency between observations due to the multiplicity of implants per patient. Relevant exposure variables (p<0.10) were incorporated into a multiple logistic regression model at patient and implant level to obtain adjusted ORs. The SPPS version 21.0 statistical package (SPSS Inc., Chicago, IL, USA) was used throughout. The level of significance was 5% (α = 0.05).

ELIGIBILITY:
Inclusion Criteria

* Males or females ≥ 18 years of age.
* One or more dental implants with an implant-supported fixed restoration.
* A minimum of one year elapsed from implant-supported restoration delivery.
* Partially edentulous patients with more than 20 teeth in the mouth.

Exclusion Criteria:

* Inaccuracy in recording peri-implant parameters due to prosthesis design.
* Implant cemented-retained prosthesis.
* Patients previously treated for peri-implantitis.
* Patients taking medications known to modify bone metabolism or with established degenerative diseases of bone (hyperparathyroidism, osteoporosis).
* Patients who had taken antibiotics, nonsteroidal antiinflammatory drugs or corticosteroids for more than two weeks in the three months before the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 years old visiting the Postgraduate Periodontology Clinic of the Faculty of Dentistry of the Universitat Internacional de Catalunya (Barcelona, Spain) from January 2018 to December 2019 were consecutively enrolled for caries exploration and dental implant condition assessment.
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of dental caries and peri-implant disease | Through the study completion, an average of 2 years
  Expressed as percentages and absolute frequencies (% and n)

SECONDARY OUTCOMES:
Mediterranean Diet adherence | Through the study completion, an average of 2 years
  This outcome was assessed by means of a questionnaire and a score. The scale score were categorised as low adherence (more or equal to 5), medium adherence (more than 5 and less or equal to 9) and high adherence (higher than >10)
Sugar consumption | Through the study completion, an average of 2 years
  Patients sugar consumption assessed dichotomously (yes/no). Sugar consumers were also asked about their level of sugar intake (low, medium, high).
Peri-implant parameters (Probing pocket depth, keratinised mucosa) | Through the study completion, an average of 2 years
  Expressed as millimetres (quantitative variables) measured at 6 sites per implant
Peri-implant parameters (Bleeding on probing, suppuration) | Through the study completion, an average of 2 years
  Assessed dichotomously (yes/no) at 6 sites per implant
Body Mass Index (BMI) | Through the study completion, an average of 2 years
  Recorded as weight (kg)/ height (m)2 and classified as underweight, normal weight, overweight or obesity.
Diabetes mellitus | Through the study completion, an average of 2 years
  presence or absence. In the case of diabetic patients, glycemic control was assessed on the basis of a previous blood test.
Nutrition or vitamin deficiency | Through the study completion, an average of 2 years
  Recorded as presence or absence
Oral dryness | Through the study completion, an average of 2 years
  Patient perception of dry mouth (presence or absence).
Educational level (EL) | Through the study completion, an average of 2 years
  primary and secondary or professional and university
Oral hygiene measures | Through the study completion, an average of 2 years
  Frequency of teeth brushing and interproximal hygiene.
Supportive periodontal treatment | Through the study completion, an average of 2 years
  Regular (≥ 2 times/year) or irregular (< 2 times/year).
Cause of tooth loss | Through the study completion, an average of 2 years
  Assessed as caries, mobility, caries and mobility, and trauma/fracture.
History of periodontitis | Through the study completion, an average of 2 years
  Assessed radiographically by the presence or absence of bone loss.
Implant position | Through the study completion, an average of 2 years
  Assessed as anterior or posterior, maxilla or mandible
Interproximal untreated caries or fillings adjacent to implants | Through the study completion, an average of 2 years
  Assessed as yes/no. If these conditions were present, their location was recorded (mesial, distal or both)
Radiographic bone level | Through the study completion, an average of 2 years
  Assessed in milimmeters at mesial and distal aspects
Age | Through the study completion, an average of 2 years
  Expressed as years
Gender | Through the study completion, an average of 2 years
  Expressed as male or female
Smoking habit | Through the study completion, an average of 2 years
  Expressed as smoker, non-smoker or ex-smoker. In the case of smokers, the total amount of cigarettes per day was categorized as < 10 or less or equal to 10 cigarettes per day.
Systemic diseases | Through the study completion, an average of 2 years
  Assessed as yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, Dr, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S313-S318. doi: 10.1002/JPER.17-0739. PMID 29926955
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215